CLINICAL TRIAL: NCT02527655
Title: Shape the Path: Targeting the Health and Mobility of Older Men Through Key Community Partnerships -- The Men on the Move Study
Brief Title: The Men on the Move Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Centre for Hip Health and Mobility (Unknown)
Responsible Party: Principal Investigator, Dawn C. Mackey, Assistant Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STP-MOTM; TE1-138295 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2015-07-29; First posted 2015-08-19 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-02

CONDITIONS: Physical Inactivity; Mobility Limitation; Older Men
MeSH Terms: conditions — Sedentary Behavior; Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Choice-Based Physical Activity and Active Transportation (Experimental): Participants will meet one-on-one with an activity coach to develop a choice-based physical activity and active transportation plan based on their interest, abilities, and resources; attend group-based motivational meetings; and receive ongoing support and encouragement for physical activity and active transportation (e.g., telephone-assisted support, community centre and transit passes).
  Interventions: Behavioral: Choice-Based Physical Activity and Active Transportation
- Wait-List Control (No Intervention): Participants will be offered the Choice-Based Physical Activity and Active Transportation intervention after the experimental arm has completed the study.

INTERVENTIONS:
Behavioral: Choice-Based Physical Activity and Active Transportation
  Arms: Choice-Based Physical Activity and Active Transportation

SUMMARY:
The Men on the Move Study is a randomized, controlled, feasibility study designed to address the health problem of physical inactivity in older men.

DETAILED DESCRIPTION:
Men on the Move is a randomized, controlled, feasibility study to provide preliminary evidence of feasibility and efficacy for promoting mobility through the uptake of physical activity among men aged 65 years and older who are physically inactive. Specifically, Men on the Move will evaluate the effects of a choice-based physical activity model paired with an active transportation model. The choice-based physical activity model encourages older men to use existing community-based resources to create and implement actions plans for physical activity. It also provides ongoing face-to-face and telephone-based support from trained activity coaches. The active transportation model provides transit passes and active travel planning to promote use of transit and walking to destinations of interest. The feasibility of delivering the intervention will be assessed. Accelerometry and travel diaries will be used to measure the effects of the intervention on physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age and older;
2. identify as a man;
3. English speaking; and
4. demonstrate readiness for physical activity (by the PAR-Q+ questionnaire or a letter of recommendation from their physician)

Exclusion Criteria:

1. participated in any strength training in the past 3 months;
2. participated in any aerobic exercise class in the past 3 months;
3. live in a nursing home or assisted living facility; or
4. have plans to be out of town for more than 7 days during the 12-week intervention period.

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of participant recruitment and retention | 12 weeks
  Number of study participants recruited and retained for the 12-week study

SECONDARY OUTCOMES:
Change from baseline in physical activity as measured by accelerometry at 12 weeks | Baseline and 12 weeks
  Minutes/day
Change from baseline in daily steps as measured by accelerometry at 12 weeks | Baseline and 12 weeks
  steps/day
Change from baseline in physical activity as measured by the CHAMPS questionnaire score at 12 weeks | Baseline and 12 weeks
Change from baseline in active transportation as measured by travel diaries at 12 weeks | Baseline and 12 weeks
  Trip rates (overall, by walking, by transit)
Change from baseline in mobility as measured by the Short Physical Performance Battery (SPPB) score at 12 weeks | Baseline and 12 weeks
Change from baseline in mobility as measured by the Life-Space Assessment score at 12 weeks | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dawn C Mackey, PhD, Principal Investigator — Simon Fraser University; Heather A McKay, PhD, Principal Investigator — University of British Columbia; Meghan Winters, PhD, Principal Investigator — Simon Fraser University; Joanie Sims-Gould, PhD, Principal Investigator — University of British Columbia; Christiane Hoppmann, PhD, Principal Investigator — University of British Columbia; Alison Phinney, PhD, Principal Investigator — University of British Columbia; Karim Khan, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Centre for Hip Health and Mobility, Vancouver, British Columbia, Canada